CLINICAL TRIAL: NCT00616577
Title: Preemptive Analgesia in Children Using Caudal Epidural Ropivacaine: A Prospective, Randomized, Double-blinded, Controlled Study
Brief Title: Preemptive Analgesia in Children Using Caudal Epidural Ropivacaine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is no longer here.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 57235
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Results first posted 2015-04-08 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Inguinal Herniorrhaphy; Orchiopexy
Keywords: Caudal Epidural Ropivacaine
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group CB (Experimental): Subjects in this arm will receive caudal ropivacaine 0.25% at a dose of 1ml/kg (maximum 15ml) with 1:200,000 epinephrine after induction of general anesthesia prior to surgical incision.
  Interventions: Drug: Ropivacaine
- Group CA (Active Comparator): Group CA (Caudal After-control group) will receive caudal ropivacaine 0.25% at a dose of 1ml/kg (maximum 15ml) with 1:200,000 epinephrine after completion of surgery but before emergence from anesthesia.
  Interventions: Drug: Ropivacaine
- Group LIA (Active Comparator): Group LIA (Local Infiltration After-control group) will receive local infiltration of ropivacaine 0.25% up to 1ml/kg (maximum 15ml) around the surgery site at the conclusion of surgery but before emergence from anesthesia.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — caudal ropivacaine 0.25% at a dose of 1ml/kg (maximum 15ml) with 1:200,000 epinephrine
  Arms: Group CB
Drug: Ropivacaine — caudal ropivacaine 0.25% at a dose of 1ml/kg (maximum 15ml) with 1:200,000 epinephrine
  Arms: Group CA
Drug: Ropivacaine — local infiltration of ropivacaine 0.25% up to 1ml/kg (maximum 15ml) around the surgery site
  Arms: Group LIA

SUMMARY:
Caudal epidural analgesia (caudal block) is used in standard pediatric anesthesia practice. It has been shown to be effective in managing postoperative pain in children undergoing abdominal and infraumbilical surgery (Tobias et al 1994). Furthermore, studies have shown that children receiving caudal blocks have secondary benefits such as lower narcotic and anesthetic requirements, more rapid awakening from general anesthesia, decreased time to discharge home, and fewer pain-related behaviors postoperatively (Conroy et al 1993, Tobias et al 1995, Tobias 1996).

This proposed study involves the use of a caudal block in children undergoing elective inguinal herniorrhaphy or orchiopexy to evaluate the role of preemptive analgesia in pediatric pain management. We hypothesize that by inhibiting peripheral pain receptors with a caudal block before the onset of a painful stimulus, we can decrease central nervous system sensitization and reduce postoperative analgesic requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 years or younger.
* Weight 33 kg or less.
* Scheduled for elective inguinal herniorrhaphy or orchiopexy.
* American Society of Anesthesiologists Class 1, 2 or 3.

Exclusion Criteria:

* Age over 2 years.
* Weight over 33 kg.
* Allergy to ropivacaine.
* Usual contraindications to caudal anesthesia (patient refusal, skeletal or spinal cord anomaly, coagulopathy, infection at insertion site, ongoing bacteremia)

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2007-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Lee, M.D., Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: IRB annual renewal indicates 26 participants Resident on the project indicates only 22 started the study.
Period: Overall Study
Arm/Group | Group CB | Group CA | Group LIA
Started | 6 | 9 | 7
Completed | 6 | 9 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: PI left institution and records cannot be located
Groups:
- Total: Total of all reporting groups
Arm/Group | Group CB | Group CA | Group LIA | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Usage of Pain Medications
Time Frame: Over 24 hours
Population: PI left institution and records cannot be located.
Arm/Group | Group CB | Group CA | Group LIA
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: Cannot verify AE occurrence. PI has left the institution and records cannot be located.
Arm/Group | Group CB | Group CA | Group LIA
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes